CLINICAL TRIAL: NCT05060653
Title: Stereotactic Body Radiotherapy Followed by Surgical Stabilization for Patients With Unstable Spinal Metastases: Cohort Study According to the IDEAL Recommendations
Brief Title: Stereotactic Body Radiotherapy Followed by Surgical Stabilization in Spinal Metastases
Acronym: BLEND-II
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Alternative study was set up
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, J.J. Verlaan, Principal investigator, UMC Utrecht
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL76750.041.21
Record Dates: First submitted 2021-08-06; First posted 2021-09-29 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Spinal Neoplasms; Neoplasm Metastasis; Radiosurgery; Surgery
MeSH Terms: conditions — Spinal Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SBRT followed by surgical stabilization within 48 hours (Experimental): SBRT and surgical stabilization will be performed within a 24 to 48-hour time window instead of today's standard of care of two weeks between surgical stabilization and conventional radiotherapy.
  Interventions: Other: SBRT followed by surgical stabilization within 24-48 hours

INTERVENTIONS:
Other: SBRT followed by surgical stabilization within 24-48 hours — In a first step, patients will undergo SBRT with active sparing of the surgical site. Patients will receive high dose, single to few fractions radiotherapy consisting of a boost to the metastases exclusively. The bony compartment containing the metastatic lesion will receive an elective dose in order to treat subclinical disease. Treatment planning is performed on the pre-treatment CT and MRI data in radiotherapy position that are mutually registered to yield information on all relevant structures for planning. Dose constraints are set for the organ at risks based on institution specific guidelines. All patients will be treated with on online position verification protocol based on institution specific guidelines. Hereafter, surgical intervention will be performed to the standard of care.

SUMMARY:
The aim of this study is to assess pain response after combining stereotactic body radiotherapy (SBRT) and pedicle screw fixation in a 48-hour window for the treatment of painful unstable metastases of the thoracic and/or lumbar spine.

DETAILED DESCRIPTION:
Rationale Sixty-five percent of cancer patients with terminal illness have bone metastases, with debilitating pain often as the severe consequence. The spine is the most common location for bone metastases. Standard treatment of unstable vertebral metastases consists of stabilizing surgery, followed by external beam radiotherapy after two weeks. Although this approach is effective in 60-70% of patients, it is has several downsides. Firstly, because of the two weeks interval between surgery and external beam radiotherapy, necessary for sufficient wound healing, it takes time before radiotherapy-induced pain relief is achieved. Moreover, the surgical implants used cause scatter artifacts on planning computed tomography images which prohibits high-resolution imaging and accurate targeting of the lesion. Multiple hospital visits (ranging from 1 to 10) are needed for administration of external beam irradiation, and in about 30-40% of patients no adequate pain response is achieved. An alternative treatment strategy, which would lead to faster pain relief in a higher proportion of patients with less hospital visits, would be highly desirable from the patient's perspective. Secondly, this strategy delays the start of systemic therapy.

Objective The main outcome of this study is pain response 4 weeks after start of the treatment.

Study design Prospective cohort study nested within the PRESENT cohort being a phase 2b study according to the IDEAL recommendations

Study population All patients, male and female, with impending spinal instability requiring surgical intervention and radiotherapy at the University Medical Center Utrecht

Intervention The combined treatment of stereotactic body radiotherapy and pedicle screw fixation in a 24 to 48-hour window for the treatment of painful unstable metastases of the cervical, thoracic and/or lumbar spine.

Main study parameters/endpoints The main outcome of this study is pain response after 4 weeks

Nature and extent of the burden and risks associated with participation, benefit and group relatedness In the preceding BLEND First-in-man study, the investigators have observed no Serious Adverse Events after a median follow-up of 13 months demonstrating the safety and feasibility of this approach.

ELIGIBILITY:
Inclusion Criteria:

* Participation in PRESENT cohort
* Painful radiosensitive metastases from solid tumors in the cervical, thoracic or lumbar spine needing surgical stabilization
* Histologic proof of malignancy or radiographic/clinical characteristics indicating malignancy beyond reasonable doubt
* Radiographic evidence of spinal metastases
* Fit for (radio)surgery
* Age > 18 years at the time of given informed consent in the PRESENT cohort.
* Written informed consent

Exclusion Criteria:

* SBRT cannot be delivered, e.g. in patients who cannot lie on the treatment table because of pain
* Surgery cannot be performed, e.g. in patients with multiple spinal metastases that cannot be bridged
* Previous surgery or radiotherapy to index lesion
* Neurological deficits (ASIA C, B or A)
* Partial neurological deficits (ASIA D) with rapid progression (hours to days)
* Non-ambulatory patients
* Patient in hospice or with < 3 months life expectancy
* Medically inoperable or patient refused surgery
* Radiosensitizing systemic treatment that cannot reasonably be stopped (for example immunotherapy and EGFR inhibitors)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Pain response | 4 weeks
  Pain response is defined as a decrease in initial worst pain score by at least 2 points on a Numeric Rating Scale (NRS) of 10 at the treated site, without increase in analgesic use, or an analgesic decrease of at least 25% without an increase in pain score

SECONDARY OUTCOMES:
Duration of pain relief | Through hospital stay, an average of 3 days
  Duration of pain relief, as measured by the Brief Pain Inventory (BPI)
Length of hospital stay | Through hospital stay, an average of 3 days
  Length of hospital stay in days
30-day mortality | 30 days
  Mortality after 30 days
Neurological status | Through hospital stay, an average of 3 days
  American Spinal Injury Association (ASIA) scale as measured by physical examination of neurologists or trained ASIA physician
Neurological deterioration | Through hospital stay, an average of 3 days
  Defined as a deterioration on the American Spinal Injury Association (ASIA) scale of more than one level
Adverse events | Through hospital stay, an average of 3 days
  Adverse events will be scored using a SAVES form

CONTACTS AND LOCATIONS:
Overall Officials: Jorrit-Jan Verlaan, MD, PhD, Principal Investigator — UMC Utrecht
Locations (1):
- UMC Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No
IPD may be shared when requested through the principal investigator